CLINICAL TRIAL: NCT01660711
Title: A Pilot Study of Neoadjuvant and Adjuvant mFOLFIRINOX in Localized, Resectable Pancreatic Adenocarcinoma
Brief Title: A Pilot Study of Pre- and Post-surgery Chemotherapy With mFOLFIRINOX in Localized, Resectable Pancreatic Adenocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Endeavor Health (Other)
Collaborators: University of Chicago (Other)
Responsible Party: Principal Investigator, Robert de W Marsh MD, Section Chief Gastrointestinal Oncology, Clinical Professor University of Chicago, Endeavor Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EH12-267
Record Dates: First submitted 2012-08-03; First posted 2012-08-09 (Estimated); Results first posted 2021-11-08 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-11

CONDITIONS: Pancreatic Adenocarcinoma
Keywords: neoadjuvant; chemotherapy; resectable; adjuvant; pancreas; cancer; adenocarcinoma; surgery
MeSH Terms: conditions — Neoplasms; Adenocarcinoma | interventions — Fluorouracil; Leucovorin; Irinotecan; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- FOLFIRINOX chemotherapy (Experimental): 5FU 2400 mg/m2 IV over 48 hours Irinotecan 180 mg/m2 IV day 1 Oxaliplatin 85 mg/m2 IV day 1 Leucovorin 400 mg/m2 IV day 1
  Cycles administered every 14 days for 4 cycles before and 4 cycles after surgery.
  Interventions: Drug: 5 Fluorouracil; Drug: Leucovorin; Drug: Irinotecan; Drug: Oxaliplatin

INTERVENTIONS:
Drug: 5 Fluorouracil — 2400 mg/m2 by continuous intravenous infusion over 46 hours
  Other Names: Adrucil,5FU
Drug: Leucovorin — 400 mg/m2 by IV infusion over 2 hours
  Other Names: Folinic acid, Wellcovorin, citrovorum factor
Drug: Irinotecan — 180 mg/m² IV infusion on Day 1 over 90-120 minutes (infusion via a Y connector during the infusion of leucovorin)
  Other Names: camptosar, CPT11
Drug: Oxaliplatin — 85 mg/m² IV infusion on Day 1 over 2 hours
  Other Names: Eloxatin,

SUMMARY:
The purpose of the study is to demonstrate that it is possible to administer chemotherapy prior to and following surgery for pancreatic cancer which is considered operable. The chemotherapy chosen is that which has been shown to be the most effective in treating metastatic disease, and the goal is both to investigate whether this is tolerable and also to investigate the efficacy of this approach in terms of disease response and survival.

DETAILED DESCRIPTION:
Pancreatic ductal adenocarcinoma is a highly lethal disease. It is estimated that in 2010 there were approximately 43,140 new cases in the United States and 36,800 deaths which ranks fourth among cancer related deaths . At diagnosis, roughly 17,000 of the initial 43,000 patients have disease which appears to be localized to the pancreatic bed, but unfortunately, only a minority of these patients (15-20%) are immediately operable (on imaging studies their disease appears to be both localized to the pancreas and technically resectable with clear margins, and at surgery no unexpected findings preclude an R0 resection ). It should be noted that of those patients deemed immediately operable on clinical grounds, between 20 and 57% are found to have inoperable disease on exploration depending on the series and on the extent and nature of preoperative staging. The majority of patients have locally advanced, borderline resectable or unresectable disease owing to involvement of critical structures, most particularly sentinel blood vessels such as the SMA, celiac axis, hepatic artery, SMV, or portal vein. Furthermore, despite recent advances in systemic therapy, even those fortunate few able to undergo immediate surgery remain largely incurable, with a five year survival of slightly less than 20%.

The current standard of care for adjuvant therapy in resectable pancreatic cancer is based on the CONKO-001 study which randomized patients to 6 cycles of postoperative adjuvant therapy with gemcitabine versus observation alone. Results favored adjuvant gemcitabine in both disease free survival (13.4 vs 6.9 months, p<0.001) and overall survival (24.2 months vs 20.5 months p=0.02) strongly supporting the use of adjuvant gemcitabine in the setting of both R0 and R1 resections. An RTOG study - 97-04 - concluded that gemcitabine was probably superior to 5FU when used pre and postoperatively in combination with 5FU/RT, with a HR of 0.82. The role of radiation therapy in this setting remains controversial, with studies such as the GITSG trial (pro) and ESPAC 1 (con) criticized either for questionable design, outdated chemotherapy or unconventional radiation therapy. Current studies in progress examining postoperative therapy include RTOG 0848 (phase III looking at adjuvant gemcitabine versus gemcitabine plus erlotinib plus/minus chemo/RT using fluorouracil), ACOSOG Z5041 evaluating gemcitabine plus erlotinib in the pre and postoperative setting and ESPAC 4 evaluating gemcitabine versus gemcitabine plus capecitabine.

Many studies have explored the use of neoadjuvant therapy in initially resectable, borderline resectable and unresectable disease. The majority of these have been single arm, single institution phase I/II studies, and results have been mixed. Potential benefits of a neoadjuvant approach include: downstaging of disease with an increased percentage of margin negative and lymph node negative resections; no delay in systemic therapy aimed at eradicating micrometastatic disease; the detection of biologically aggressive tumors, as evidenced by early progression/metastases during this phase of therapy, thereby avoiding inappropriate surgery; and the greater likelihood of completing all intended therapy as opposed to postoperative treatment, where fully 22 - 35% of patients do not complete their intended program.

A comprehensive meta-analysis and systematic review of neoadjuvant therapy in both resectable and unresectable pancreatic cancer has recently been published. The conclusion reached in resectable patients was that resection frequency and survival following neoadjuvant therapy was similar to that in patients undergoing primary resection followed by adjuvant therapy. In patients with initially unresectable disease, fully one third had resectable tumors following neoadjuvant therapy with survival comparable to initially resectable patients. In aggregate, these observations indicate that a neoadjuvant approach is feasible and effective, and that this sequence does not compromise resectability or survival, even in those patients with the best prognosis.

With respect to specific studies in resectable disease, investigators at MD Anderson Cancer Center have published their most recent results. In their first study, 86 patients with resectable disease in the head of the pancreas received radiation therapy (30 Gy in 10 fractions over 2 weeks) plus 7 weekly infusions of gemcitabine at 400 mg/m2/week. 85% of these patients were taken to surgery and 74% were able to undergo the intended pancreaticoduodenectomy. Median survival for patients whose disease was resected was 34 months, but it was only 7 months for those whose disease could not be resected. In a second study of patients with resectable adenocarcinoma of the pancreatic head, 90 patients were enrolled with the goal of administering chemotherapy alone for eight weeks, using gemcitabine and cisplatin, followed by combined low dose gemcitabine and radiation therapy (30 Gy in 10 fractions). Ultimately, 79 (88%) patients completed the full course of preoperative therapy and 62 of these (78%) patients were taken to surgery. 52 (66%) had their disease resected with a median survival of 31 months for those who had surgery, versus 10.5 months for those who did not. They concluded that initial combination chemotherapy with gemcitabine and cisplatin followed by chemotherapy/RT did not improve on the results achieved with chemotherapy/RT alone. This result is perhaps not surprising as gemcitabine, both alone and in doublet combinations, has simply not been active enough to materially impact on the outcome of this disease. Interestingly, the longer preoperative interval did not result in local tumor progression.

These findings are similar to those of other major centers reporting studies of neoadjuvant gemcitabine based chemoradiation for potentially resectable disease, and suggest that this is a valid strategy for further study in this setting.

Recently, investigators in Europe reported their results with a novel combination of docetaxel 30 mg/m2 weekly and RT of 45 Gy in 34 patients with resectable disease. 32% had progression, 59% stable disease and 9% partial remission. 50% of the original cohort had pancreaticoduodenectomy with 100% R0 resection and a median survival of 32 months. The numbers are small and the overall resection rate disappointingly low, but the R0 resection rate and median survival for those resected is equivalent to patients receiving gemcitabine based regimens.

In locally advanced, unresectable disease, results have recently been reported from Austria with neoadjuvant gemcitabine/oxaliplatin without RT (39% of patients undergoing resection of disease with 69% R0 and 22 months median survival), Italy with neoadjuvant PEFG/PEXG (cisplatin, epirubicin, 5-fluorouracil (F)/capecitabine (X), gemcitabine) or PDXG (docetaxel substituting for epirubicin) followed by RT plus X, F or G (14% resected with median survival 16.2 months)and Japan with neoadjuvant gemcitabine 1000 mg/m2/wk and RT 50 Gy in T3 disease followed by postoperative 5FU liver perfusion (82% of patients with disease resected, 43% 5 year survival). In each of these studies, there is a mixture of borderline resectable and unresectable disease with the result that the interpretation of outcomes is problematic. However, it is clear that a neoadjuvant approach is feasible and active.

It is clear from an examination of the NCI CTEP database that the neoadjuvant approach has been widely embraced for future study. More than 40 active protocols are listed, including the following select few: a UVA study of hypofractionated RT plus chronomodulated capecitabine in resectable and borderline resectable disease; a UT Southwestern phase I study of SBRT or SBRT plus gemcitabine; an Emory phase I study of FOLFIRINOX and SBRT; a Fred Hutchinson study of GTX and oxaliplatin with IMRT and adjuvant gemcitabine; a UF phase II study of risk adapted gemcitabine plus abraxane; a European randomized phase II study of gemcitabine plus oxaliplatin pre and gemcitabine postoperatively versus gemcitabine postoperatively only; a Memorial Sloan Kettering phase II study of gemcitabine plus oxaliplatin preoperatively plus gemcitabine postoperatively; and an ACOSOG study of gemcitabine plus erlotinib pre and postoperatively.

Looking to the future there have been a number of recent innovations in chemotherapy. In an ongoing effort to discover non-gemcitabine based chemotherapy for those who have progressed on gemcitabine, and also a new regimen with more efficacy than those currently used in patients with pancreatic cancer, the combination of 5FU, leucovorin, oxaliplatin and irinotecan has been tested. This combination was initially studied in colorectal cancer, in a regimen known as FOLFOXIRI. It was established that this combination was both tolerable and effective in this setting. Subsequently, the regimen was modified slightly to the current FOLFIRINOX format (oxaliplatin 85mg/m2, irinotecan 180 mg/m2, leucovorin 400 mg/m2 , 5FU 400 mg/m2 on day 1, then 5FU 2400 mg/m2 as a 46 hour continuous infusion) and tested in a phase II study in pancreatic cancer. 47 chemotherapy-naïve patients with metastatic disease were enrolled and 46 were treated. Confirmed response rate was 26% with 4% complete responses. Median time to progression was 8.2 months and median overall survival was 10.2 months. Grade 3/4 toxicities included neutropenia (52%), nausea (20%), vomiting (17%), diarrhea (15%), and neuropathy (15%). No toxic death occurred. FOLFIRINOX was then tested after failure of previous gemcitabine therapy in metastatic disease and was deemed to be promising. 13 patients were treated, with 9 evaluable for response - 6 had stable disease with a mean time to progression of 6.6 months, and 3 progressed.

As a consequence of the previously mentioned phase II study in chemo-naïve patients, a randomized phase II/phase III study comparing gemcitabine (G) to FOLFIRINOX (F) as first line treatment of metastatic pancreatic cancer was conducted. This study was terminated prematurely by the study IDMC as it was determined that additional patient accrual would not add to the statistical power of the study. 342 patients were accrued with roughly one third of the primary disease involving the head of the pancreas. Overall objective response rate was 32% for F versus 9.4% for G. PFS was 6.4 months versus 3.4 months and overall survival 11.1 months versus 6.8 months, all in favor of F.

The overall survival rate of 11.1 months is the best result achieved thus far in a randomized phase III study of chemotherapy in metastatic pancreatic cancer. Notable toxicities of at least grade III/IV, which were all worse with F, were neutropenia (45.7 vs 18.7%), febrile neutropenia (5.4 vs 0.6%), fatigue (23.7 vs 14.2%), vomiting (14.5 vs 4.7%) and diarrhea (12.7 vs 1.2%). These results indicate that this is a notably active regimen with an encouraging response rate. However, the potential toxicities are significant, and it is a regimen that should be offered only to patients with ECOG 0-1 performance status and excellent supportive care. In this regard, in an attempt to ameliorate these toxicities, modifications to the published regimen have already been proposed by the French group and others. In their forthcoming study of FOLFIRINOX in the adjuvant setting, the French will omit the bolus of 5FU which contributes significantly to the myelosuppression but which is thought to have minimal impact on the therapeutic efficacy. In addition, most physicians now incorporate the routine use of neulasta with each treatment cycle. This study will similarly incorporate these modifications and the regimen will be named mFOLFIRINOX.

Thus, in the context of perioperative therapy, we have identified a regimen - FOLFIRINOX - with the best results to date in the treatment of metastatic disease and by inference, promise of improved outcome in those patients with resectable disease. If successful, this has the potential to improve DFS and overall survival (until now no better than 15-20% at 5 years) in these patients, and may establish a new paradigm for future studies.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic diagnosis of adenocarcinoma of the pancreas.
* Resectable primary tumor of the head, body or tail of the pancreas defined as a visible mass in the pancreas and:
* No extrapancreatic disease
* A patent superior mesenteric (SMV)- portal vein (PV) confluence (assuming the technical ability to resect and reconstruct this venous confluence if needed)
* A definable tissue plane between the tumor and regional arterial structures including the celiac axis, common hepatic artery, and SMA.
* Confirmation of resectability by surgical oncology consultation.
* Presentation at a multidisciplinary conference at either University of Chicago or NorthShore University
* No previous therapy for pancreatic cancer
* Short removable metal stents rather than plastic stents are preferred but not required for palliation of initial obstructive jaundice
* Karnofsky performance status 80 or better
* Age > 21 years
* No currently active second malignancy
* No CVA within 6 months, no MI within 6 months
* The effects of mFOLFIRINOX on the developing human fetus are unknown. For this reason and because chemotherapy agents as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Negative pregnancy test in females of reproductive age
* Life expectancy of greater than 3 months.
* Anticoagulation is permitted but patients may only be on lovenox for this purpose.
* Patients must have normal organ and marrow function as defined below:

  * absolute neutrophil count >1,500/mcL
  * platelets >100,000/mcL
  * total bilirubin <1.5X upper limits of normal
  * AST(SGOT)/ALT(SGPT) <2.5 X institutional upper limit of normal
  * creatinine within normal institutional limits OR
  * creatinine clearance >60 mL/min/ per Cockcroft-Gault equation for patients with creatinine levels above institutional normal.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients who have had previous chemotherapy or radiotherapy for pancreatic adenocarcinoma prior to entering the study.
* Pathologic subtypes other than pure adenocarcinoma; acinar cell carcinoma, squamous cell carcinoma, spindle cell carcinoma, neuroendocrine cancer, and mixed types are not eligible.
* Patients who are receiving any investigational agents.
* Patients with borderline resectable, locally advanced or metastatic disease.
* History of allergic reactions attributed to 5FU, leucovorin, irinotecan or oxaliplatin or to compounds of similar chemical or biologic composition.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, active liver disease including viral or non-viral hepatitis and cirrhosis, chronic diarrhea or inflammatory disease of the colon or rectum, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study. mFOLFIRINOX is a regimen containing more than one chemotherapy agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with FOLFIRINOX, breastfeeding should be discontinued if the mother is treated with these agents. These potential risks may also apply to other agents used in this study.
* HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with mFOLFIRINOX. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.
* Currently active second malignancy other than non-melanoma skin cancer or carcinoma in-situ of the cervix. Patients are not considered to have a "currently active" malignancy if they have completed therapy and have no evidence of recurrence for at least 5 years.
* Pre-existing neuropathy greater than grade 1.
* Anticoagulants other than low molecular weight heparin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2012-07; Primary Completion 2018-08-22 (Actual); Study Completion 2018-08-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- NorthShore University HealthSystem, Evanston, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- FOLFIRINOX Chemotherapy: 5FU 2400 mg/m2 IV over 48 hours Irinotecan 180 mg/m2 IV day 1 Oxaliplatin 85 mg/m2 IV day 1 Leucovorin 400 mg/m2 IV day 1
  Cycles administered every 14 days for 4 cycles before and 4 cycles after surgery.
  5 Fluorouracil: 2400 mg/m2 by continuous intravenous infusion over 46 hours
  Leucovorin: 400 mg/m2 by IV infusion over 2 hours
  Irinotecan: 180 mg/m² IV infusion on Day 1 over 90-120 minutes (infusion via a Y connector during the infusion of leucovorin)
  Oxaliplatin: 85 mg/m² IV infusion on Day 1 over 2 hours
Period: Overall Study
Arm/Group | FOLFIRINOX Chemotherapy
Started | 22
Completed | 14
Not Completed | 8
Not completed — Adverse Event | 7
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- FOLFIRINOX Chemotherapy: All participants.
Arm/Group | FOLFIRINOX Chemotherapy
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants] — Population: 1 person registered was ineligible and did not participate.
  Participants
    <=18 years | 0
    Between 18 and 65 years | 17
    >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 13
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Percentage Able to Complete Full Course of Preoperative Chemotherapy
Description: The percentage of participants able to complete the full course of preoperative chemotherapy and undergo a resection. This will be the primary determinant of success for this pilot study. - Early withdrawals due to toxicity, disease progression, or intercurrent illness will be considered failures.
Time Frame: Following completion of all planned therapy, an expected average of 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | FOLFIRINOX Chemotherapy
Number analyzed (Participants) | 22
Participants | 22

2. Secondary Outcome: Percentage Able to Complete Full Course of Therapy
Description: The percentage of participants able to complete the full course of therapy, including preoperative chemotherapy, surgical resection and postoperative chemotherapy.
Time Frame: On completion of all planned therapy, an expected average of 8 months
Measure: Count of Participants; unit: Participants
Arm/Group | FOLFIRINOX Chemotherapy
Number analyzed (Participants) | 22
Participants | 14

3. Other Pre Specified Outcome: Treatment Related Toxicity
Description: Treatment related toxicity and other adverse events (AEs) during Toxicity of preoperative and postoperative therapy and the safety of this approach.
Time Frame: 1 year
Reporting Status: Not Posted

4. Other Pre Specified Outcome: R0 Resection Rate
Description: Assessment of the percentage of patients able to have an R0 resection following preoperative chemotherapy.
Time Frame: 3 months
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Progression-free and Overall Survival
Description: Assessment of progression-free survival and overall survival from the start of study treatment.
Time Frame: 5 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 2 years
Groups:
- FOLFIRINOX Chemotherapy: FOLFIRINOX chemotherapy in all participants.
Arm/Group | FOLFIRINOX Chemotherapy
All-Cause Mortality (participants affected / at risk) | 2/22
Serious Adverse Events (participants affected / at risk) | 14/22
Other Adverse Events (participants affected / at risk) | 0/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FOLFIRINOX Chemotherapy (N=22)
Diarrhea (Gastrointestinal disorders) | 4 (4)
neutropenia (Blood and lymphatic system disorders) | 1
anorexia (Gastrointestinal disorders) | 5
Hyperglycemia (Endocrine disorders) | 2
Hypokalemia (Renal and urinary disorders) | 1
Fatigue (General disorders) | 3
peripheral neuropathy (Nervous system disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-05-13): https://cdn.clinicaltrials.gov/large-docs/11/NCT01660711/Prot_SAP_000.pdf